CLINICAL TRIAL: NCT04823182
Title: Study of HEarT DiseAse and ImmuNiTy After COVID-19 in Ireland
Acronym: SETANTA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cardiovascular Research Institute Dublin (Other)
Responsible Party: Sponsor
Other Study IDs: SETANTA_Study_Protocol_V2.0
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV Infection; Covid19; Cardiomyopathies
Keywords: Cardiac Magnetic Resonance Imaging; COVID19; Cardiomyopathy
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Cases - Recent COVID-19 infection ≥ 6 weeks and ≤ 12 months before enrolment, as evidenced by positive reverse-transcriptase polymerase chain reaction (RT-PCR) SARS-CoV-2 swab
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Cardiovascular Magnetic Resonance Imaging — The Cardiac MRI protocol consists of static T2 weighted in all three planes and T2 weighted imaging with fat saturation in the short axis plane.
  Other Names: Cardiac MRI

SUMMARY:
SETANTA study will investigate the incidence of cardiac abnormalities as assessed by cardiac magnetic resonance imaging in unselected patients after acute SARS-CoV-2 infection and correlation with immunological response and biomarkers of coagulation.

DETAILED DESCRIPTION:
Approximately 100 participants from primary care will be enrolled via General Practitioner (GP) or Primary Care Centers in Dublin. A patient information sheet (PIS) will be made accessible to participants recovering from COVID-19 via their GP practice inviting the participants to contact Cardiovascular Research Institute Dublin. The participants, subject to suitability, will be invited for a site visit over two days, where upon explicit consent being granted, the Investigators will proceed with data collection. The study population includes participants who are recovering from COVID-19 in the community.

Primary Objective

To investigate the incidence of cardiac abnormalities as assessed by cardiac magnetic resonance imaging in unselected participants after acute SARS-CoV-2 infection and correlation with immunological response and biomarkers of coagulation.

Secondary Objectives

* To investigate the incidence of SARS-CoV-2 immunity and
* To investigate the extent of coagulopathy persistent after acute SARS-CoV-2 infection.

Follow-up data collection points will be at 1, 6- and 12-months including assessment of major adverse cardiovascular events (MACE) such as myocardial infarction (MI), revascularization, pulmonary embolism (PE), deep venous thromboembolism (DVT), incident heart failure and stroke. 'Patient reported outcome measures' via two quality of life (QOL) questionnaires will be administered at baseline and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. Written informed consent
3. Recent COVID-19 infection ≥ 6 weeks and ≤ 12 months before enrolment, as evidenced by positive reverse-transcriptase polymerase chain reaction (RT-PCR) SARS-CoV-2 swab

Exclusion Criteria:

1. Prior history of myocarditis or ischemic heart disease
2. General contraindications for Magnetic Resonance Imaging e.g. Magnetic Resonance unsafe pacemaker, devices, implants etc.
3. Contraindication to gadolinium (estimated glomerular filtration rate <30 ml/min)
4. Contraindication to Regadenoson, including cardiac conduction disease, asthma, seizures, pregnancy or breast-feeding
5. Inability to provide written informed consent, to fill out the safety questionnaire, or to fully cooperate with the scan and breath holds
6. Insufficient Cardiac Magnetic Resonance image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recent COVID-19 infection ≥ 6 weeks and ≤ 12 months before enrolment, as evidenced by positive reverse-transcriptase polymerase chain reaction (RT-PCR) SARS-CoV-2 swab
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-09-22 (Estimated)

PRIMARY OUTCOMES:
Left ventricular (LV) ejection fraction | Day 0
  Cardiac Magnetic Resonance finding
LV end diastolic volume | Day 0
  Cardiac Magnetic Resonance finding
Right ventricular ejection fraction | Day 0
  Cardiac Magnetic Resonance finding
Native T1, T2 | Day 0
  Cardiac Magnetic Resonance finding
Late gadolinium enhancement | Day 0
  Cardiac Magnetic Resonance finding
Pericardial abnormalities | Day 0
  Cardiac Magnetic Resonance finding

SECONDARY OUTCOMES:
Immunity parameters | Day 0
  Anti-SARS-CoV-2 total antibody testing
Markers of coagulation and endothelial cell activation | Day 0
  Including fibrinogen, D-dimer, von Willebrand factor antigen, von Willebrand factor propeptide, soluble thrombomodulin, activated protein C, and cytokine arrays

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Byrne, MB BCh PhD, Principal Investigator — CVRI Dublin at Mater Private Hospital; Roisin Colleran, MB BCh, Principal Investigator — CVRI Dublin at Mater Private Hospital
Locations (1):
- Cardiovascular Research Institute Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Colleran R, Fitzgerald S, Rai H, McGovern L, Byrne RJ, Mansur A, Cradock A, Lavery R, Bisset J, McKeogh S, Cantwell G, O'Ciardha D, Wilson H, Begossi N, Blake N, Fitzgibbon M, McNulty J, Szeplaki G, Heffernan E, Hannan M, O'Donnell JS, Byrne RA. Symptom burden, coagulopathy and heart disease after acute SARS-CoV-2 infection in primary practice. Sci Rep. 2024 Sep 11;14(1):21229. doi: 10.1038/s41598-024-71535-8. PMID 39261512